CLINICAL TRIAL: NCT02279186
Title: Effectiveness of Intravenous Tranexamic Acid in Reducing Blood Loss During and After Cesarean Section ,A Randomized Clinical Trial .
Brief Title: Effectiveness of Intravenous Tranexamic Acid in Reducing Blood Loss During and After Cesarean Section
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams Maternity Hospital (Other)
Responsible Party: Principal Investigator, Mahmoud Mostafa Abdellah Mostafa, Effectiveness of Intravenous Tranexamic Acid in Reducing Blood Loss During and After Cesarean Section ,A Randomized Clinical Trial., Ain Shams Maternity Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: septemper 2014
Record Dates: First submitted 2014-10-24; First posted 2014-10-30 (Estimated); Last update posted 2014-11-04 (Estimated); Status verified 2014-11

CONDITIONS: Bleeding
MeSH Terms: conditions — Hemorrhage | interventions — Tranexamic Acid; Sodium Chloride

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- group A (Active Comparator): receiving tranexamic acid
  Interventions: Drug: Tranexamic Acid
- group B (No Intervention): does not receive tranexamic acid

INTERVENTIONS:
Drug: Tranexamic Acid — Intravenous Injection
  Other Names: in 200 ml saline
  Arms: group A

SUMMARY:
In this study, the efficacy and safety of tranexamic acid in the reducing the blood loss during and after elective LSCS will be investigated.

DETAILED DESCRIPTION:
To state the effectiveness clinically and laboratory and safety of tranexamic acid in reducing blood loss during and after the elective lower segment cesarean section.

ELIGIBILITY:
Inclusion Criteria:

* - Women undergoing caesarean delivery for various elective indications.
* Full term primiparas / multiparas.
* Singleton pregnancy being delivered by LSCS.

Exclusion Criteria:

* - Medical problems involving the heart, liver, kidney and brain .
* Blood disorders.
* Allergy to tranexamic acid.
* History of thromboembolic disorders, abnormal placentation, severe pre-eclampsia, uterine anomalies and pathology.
* Multiple pregnancy, macrosomia.
* Polyhydromnios .
* Patients requiring blood transfusion due to anemia

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2014-09; Primary Completion 2015-03 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
Amount of blood loss during cesarean section after placental delivery till end of the operation. | during and 2hours post cesarean section

SECONDARY OUTCOMES:
1.Vital signs eg:blood pressure ,heart rate ,respiratory rate during first two post operative hours . | up to 24hours postoperative
  composite
Adverse affect of tranexamic acid on mother and neonate . | first 24 hours
  eg:drug allergy ,drug interaction ,thrombotic manifestation and the number of participant .
24 hours post operative haemoglobin and haematocrit . | after 24 hours.
  composite

CONTACTS AND LOCATIONS:
Overall Officials: Amr Abdelaziz, M.D, Principal Investigator — Ain Shams Maternity Hospital
Locations (1):
- Ain Shams Maternity Hospital, Cairo, Egypt